CLINICAL TRIAL: NCT05844813
Title: Neoadjuvant Chemotherapy Combined With Targeted Treatment in High-risk Retroperitoneal Sarcoma-- A Nationwide Multicentered Prospective Controlled Study
Brief Title: Neoadjuvant Chemotherapy Combined With Targeted Treatment in High-risk Retroperitoneal Sarcoma
Acronym: NATARS
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University International Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Peking University First Hospital (Other); Shanghai Cancer Hospital, China (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jun Chen, MD, Peking University International Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUIH-RPS01; Z221100007422042 (Other Grant/Funding Number: Beijing Municipal Science & Technology Commission, Administrative Commission of Zhongguancun Science Park)
Record Dates: First submitted 2023-04-16; First posted 2023-05-06 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Retroperitoneal Sarcoma
Keywords: Retroperitoneal Sarcoma; Neoadjuvant therapy; Target therapy; Survival

STUDY DESIGN:
Intervention Model Description: It is a prospective non-randomized controlled study. After meeting the inclusion and exclusion criteria, patients will be allocated either into the Surgery-only Group or the Neoadjuvant therapy group. Patients in the surgery-only group will directly undergo surgeries after the confirmation of diagnosis through pre-operative biopsy, while in the neoadjuvant therapy group, patients will receive neoadjuvant chemotherapy combined with target treatment for three circles followed by the sarcoma resectional surgeries.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Neoadjuvant Therapy Group (Experimental): Neoadjuvant chemotherapy + Target therapy+ Radical resectional Surgery Drugs: Doxorubicin（PLD） 40mg/㎡ d1, Ifosfamide 1g/㎡ d1-5, Anlotinib10mg d1-14 Q3weeks * 3 Circles, Watch-Wait 4-6 weeks
  Interventions: Drug: Doxorubicin+Ifosfamide+Anlotinib(AI+A); Procedure: Radical Surgery
- The Surgery only Group (Active Comparator): Procedure: Radical resectional surgery
  Interventions: Procedure: Radical Surgery

INTERVENTIONS:
Drug: Doxorubicin+Ifosfamide+Anlotinib(AI+A) — Doxorubicin（PLD） 40mg/㎡ d1, Ifosfamide（I） 1g/㎡ d1-5, Anlotinib（A）10mg d1-14 Q3weeks * 3 Circles
  Arms: The Neoadjuvant Therapy Group
Procedure: Radical Surgery — Radical sarcoma resectional surgery

SUMMARY:
The goal of this clinical trial is to explore the potential survival benefits of neoadjuvant chemotherapy combined with target treatments followed by radical surgery in patients with primary high-risk/grade retroperitoneal sarcoma.

The main questions it aims to answer are:

* Whether the 1,3-year progression-free survival time(PFS) is prolonged in the neoadjuvant therapy group, compared with the surgery-only group.
* The Overall survival time in the two groups.
* The safety and tolerance in the neoadjuvant therapy group.

Participants will be allocated into two groups once they meet the inclusion criteria.

* Surgery-only Group: Patients will directly undergo surgeries after the confirmation of diagnosis through pre-operative biopsy.
* Neoadjuvant therapy group: Patients will receive the neoadjuvant chemotherapy combined with target treatment for three circles before the following sarcoma resectional surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary high-risk Retroperitoneal sarcoma(RPS) (Including Dedifferentiated liposarcoma (DDLPS), leiomyosarcoma(LMS), Undifferentiated pleomorphic sarcoma(UPS), Solitary fibrous tumor(SFT)).
* Primary localized RPS without histories of surgical resection, chemo- or radio-therapy, targeted therapy. Patients who underwent laparotomy with biopsy only will also be considered as primary cases.
* Without histories of second malignant tumors.
* In DDLPS

  * Diagnosis should be confirmed based on MDM2(Mouse double minute 2 homolog) and CDK4(Cyclin-dependent kinase 4) expression on IHC (immunohistochemistry), while MDM2 amplification in the Fish test is highly recommended.
  * All grade 2-3 DDLPS can be included.
* In LMS

  * All grades of LMS can be included.
  * Tumor size ≥10cm
* In UPS or SFT

  * All grades of UPS can be included.
  * High-risk SFT with a score ≥6 in 'Risk stratification of SFT for development of metastasis' introduced in The 5th edition of the WHO(World Health Organization) Soft tissue sarcoma classification.
* Sarcoma without protruding across the diaphragm
* Possibility of R0/R1 resection evaluated through preoperative MDT(multi-disciplinary team) discussion
* No multi-organ or system dysfunction/failure or patients with slight dysfunction of organ/system could be easily recovered
* Tolerable of chemotherapy and surgery through MDT evaluation and tests.
* American Society of Anesthesiologist (ASA) ≤3
* Fully understand the informs and consent to participate in the study.

Exclusion Criteria:

* Sarcoma confirmed originating from the GI tract, uterus, or urinal tract.
* Patients included in the study through preoperative biopsy or MDT discussion, with WDLPS, grade 1 LPS, or other types of tumors not mentioned in the Inclusion criteria evaluating through final pathological findings.
* Sarcoma protruded into the chest cavity evaluated through preoperative imaging or surgical reports.
* Metastasis confirmed pathologically or highly suspicious metastatic lesions through radiological findings, PET-CT(Positron emission tomography) is highly recommended, MDT discussion and evaluation are needed.
* Histories of administration of Anthracyclines, Ifosfamide, and targeted agents.
* Severe contradiction to surgery and chemotherapies, including persistent myelosuppression, myocardial/cerebral/pulmonary infarction, uncontrolled cardiac arrhythmia, etc within the last 6 months
* Indication of severe infection or undergoing surgeries with high-risk hemorrhages in one month.
* Persistent one or more organ or system dysfunctions, could not be recovered prior to the study.
* Female patients who are pregnant or breastfeeding or female and male patients of reproductive potential who are not willing to employ effective birth control methods.
* Patients with psychological conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
3-year Progression Free Survival(PFS) | 3 years after first patient enrolled in
  Progression free survival will be measured from the date of surgery to the date of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
1-year PFS | 1year after first patient enrolled in.
  Progression free survival will be measured from the date of surgery to the date of progression or death, whichever occurs first.
1 year Overall survival(OS) | 1year after first patient enrolled in
  OS will be measured from the date of surgery to the date of death, whatever the causes of death.
3-year OS | 3 years after first patient enrolled in
  OS will be measured from the date of surgery to the date of death, whatever the causes of death.
5-year PFS | 5 years after first patient enrolled in.
  Progression free survival will be measured from the date of surgery to the date of progression or death, whichever occurs first.
5-year OS | 5 years after first patient enrolled in
  OS will be measured from the date of surgery to the date of death, whatever the causes of death.
Safety and toxicity of neoadjuvant therapy | 1-d, 7-d after the first date of each neoadjuvant therapy session.
  Safety and toxicity will be evaluated through blood tests, echocardiography, ECG, etc.
Postoperative morbidities | 30-d, 90-d, 1-year separately after the date of surgery.
  Operative outcomes including morbidities will be collected and compared in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Chenghua Luo, MD, PhD, Study Chair — Peking University International Hospital
Locations (6):
- China (6):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Cancer Hospital, Minhang Branch, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No